CLINICAL TRIAL: NCT01404078
Title: A RCT With Factorial Design to Compare Safety and Efficacy of 2 Capsules of the Indian Polycap Versus a Single Capsule Along With or Without Oral Potassium Among Patients With Stable Cardiovascular Disease
Brief Title: Study to Compare 2 Doses of Polycap Versus Single Dose of Polycap With or Without Pottasium
Acronym: TIPSK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. John's Research Institute (Other)
Collaborators: Population Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TIPS K; CTRI/2010/091/000054 (Registry Identifier: Clinical Trials Registry of India)
Record Dates: First submitted 2011-07-24; First posted 2011-07-27 (Estimated); Results first posted 2014-12-01 (Estimated); Last update posted 2014-12-01 (Estimated); Status verified 2014-11

CONDITIONS: Ischemic Heart Disease; Ischemic Stroke; Peripheral Vascular Disease; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Myocardial Ischemia; Ischemic Stroke; Peripheral Vascular Diseases; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SD Polycap without potassium (Active Comparator): Single dose polycap without pottasium
  Interventions: Drug: Single Dose Polycap
- DD Polycap plus potassium (Experimental): Double Dose polycap with potassium
  Interventions: Drug: Double dose Polycap

INTERVENTIONS:
Drug: Single Dose Polycap — Low strength polycap contains Ace inhibitor; betablocker; thiazide diuretic; statin; aspirin
  Other Names: Polycap
  Arms: SD Polycap without potassium
Drug: Double dose Polycap — 2 Capsules of low strength polycap with 30mEq of Potassium
  Other Names: Full dose polycap
  Arms: DD Polycap plus potassium

SUMMARY:
This is a randomized double blind 2x2 factorial controlled trial to evaluate efficacy tolerability of low strength Polycap versus two doses of low strength Polycap in patients with stable cardiovascular disease in reducing blood pressure and LDL.

To evaluate the tolerability and safety of low dose potassium supplementation compared to placebo in patients with stable cardiovascular disease.

Approximately 500 patients are planned to be randomized.

DETAILED DESCRIPTION:
Mean change in blood pressure between those taking 2capsules of the polycap versus one Difference in Rates of early discontinuation between 2 capsules of polycap versus one Rates of reported adverse effects among those taking the polycap

ELIGIBILITY:
Inclusion Criteria:

1. Individuals 40 years and above, with a seated blood pressure > 130/80 mm Hg on two consecutive readings (or BP > 120/80 mm Hg in patients under treatment with 2 or more antihypertensive medication) with one of the following

   1. Coronary artery disease; previous myocardial infarction (>7 days post uncomplicated MI), or
   2. Ischemic heart disease with significant ECG changes or a positive stress test, or
   3. Stable angina or unstable angina and with documented evidence of multi-vessel (angiography or ECG or CT angiography) coronary artery disease, or
   4. PTCA or CABG Surgery >30 days before informed consent.
   5. Cerebrovascular disease; Previous Ischemic stroke or Transient Ischemic Attacks >30 days before informed consent.
   6. High risk diabetes mellitus defined as HbA1C >7.5%, with microalbuminuria or blood pressure >140/90 mm Hg.
   7. Peripheral artery disease defined as a current or prior history of: physician diagnosed intermittent claudication or vascular surgery for atherosclerotic disease or an ankle/arm systolic blood pressure ratio ≤ 0.90 in either leg at rest, or angiographic or doppler study demonstrating ≥ 70% stenosis in a noncardiac artery.
2. Those who provide informed consent and can comply with medications and follow-up visits.

Exclusion Criteria:

1. Known hypersensitivity or intolerance to any of the study medications or a clear indication for full doses of beta blockers, RAAS blockers (ACEi, ARBs, Renin inhibitors, etc.), diuretics and statins.
2. History of bleeding or having hemorrhagic stroke anytime in the past or a need for continued anticoagulation therapy.
3. Patients having indication for higher doses of aspirin or needing more than 75mg of clopidogrel daily.
4. Have significant bradycardia (heart rate <50 beats/min) or second- or third-degree heart block without a pacemaker.
5. Planned cardiac surgery or PTCA or any non-cardiac surgery <3months of eligibility assessment.
6. Heart transplant recipient.
7. Renal dysfunction defined as serum creatinine >2 mg/dL and/or serum potassium >5.0 mEq/L.
8. Patients aged >70 years, with mild renal dysfunction defined as serum creatinine >124 µmol/L (1.4 mg/dL) or eGFR <45 ml/min/1.73 m2.
9. Hepatic dysfunction, SGOT or SGPT > 3 x ULN.
10. Taking another experimental drug or within 30days of last dose of the experimental drug.
11. Peptic ulcer disease with bleed, or bleeding diathesis.
12. Bronchial asthma or Chronic Obstructive Pulmonary Disease with asthma.
13. Gout, rheumatoid arthritis or other chronic inflammatory disease requiring long-term medications with NSAIDs.
14. Any history of muscular pain, other pathology of the muscles or past history of muscular pain secondary to taking statins or fibrates.
15. Pregnancy or lactating or women of childbearing potential with inadequate contraception.
16. Inability to attend follow up visits (due to significant disability, inadequate address or contact details, subject from a far off place, psychiatric illness etc.).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 518 (Actual)
Dates: Start 2010-04; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Prem - Pais, MD, Principal Investigator — St.Johns Research Institute

REFERENCES:
- See also: Pubmed Abstract — http://www.ncbi.nlm.nih.gov/pubmed/22787067

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Hospitals in India identified potential consenting eligible subjects with a history of stable cardiovascular disease or high risk for cardiovascular disease and subjected them to an active run in with single dose and then double dose of polycap. Only patients successfully completing the active run in (>80% compliant) were randomized into the trial
Pre-assignment Details: 725 Started on Phase 1 run in low dose polycap 645 started on phase 2 run in full dose polycap Only patients who fulfilled >80% compliance to full dose polycap were randomized to the trial
Groups:
- One Dose of Low Srength Polycap: Patients in this arm will receive one dose of low strength Polycap
  Indian Polycap: Polycap contains 5 drugs at half doses Ace inhibitor; betablocker; thiazide diuretic; statin; aspirin
- Two Doses of Low Strength Polycap: Patients in this arm will receive 2 doses of low strength Polycap.
  Indian Polycap: Polycap contains 5 drugs at half doses Ace inhibitor; betablocker; thiazide diuretic; statin; aspirin
Period: Overall Study
Arm/Group | One Dose of Low Srength Polycap | Two Doses of Low Strength Polycap
Started | 261 (725 Started on Phase 1 run in low dose polycap 645 started on phase 2 run in full dose polycap) | 257 (725 Started on Phase 1 run in low dose polycap 645 started on phase 2 run in full dose polycap)
Completed | 243 | 237
Not Completed | 18 | 20

BASELINE CHARACTERISTICS:
Groups:
- Polycap Single Dose: Patients in this arm received single dose of low strength Polycap only Indian Polycap: Polycap contains 5 drugs at half doses Ace inhibitor; betablocker; thiazide diuretic; statin; aspirin
- Polycap Double Dose Plus Potassium: Patients in this arm received one dose of low strength Polycap with potassium
  Indian Polycap: Polycap contains 5 drugs at half doses Ace inhibitor; betablocker; thiazide diuretic; statin; aspirin
- Total: Total of all reporting groups
Arm/Group | Polycap Single Dose | Polycap Double Dose Plus Potassium | Total
Number analyzed (Participants) | 257 | 261 | 518
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.2 (19.4) | 57.9 (19.2) | 57.6 (19.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103 | 108 | 211
  Male | 154 | 153 | 307
Region of Enrollment [Number; unit: participants]
  India | 257 | 261 | 518

OUTCOME MEASURES:

1. Primary Outcome: BLOOD PRESSURE LIPIDS
Description: Amongst patients with cardiovascular disease or type 2 diabetes, the study aims to test the safety and efficacy of giving double dose of polycap versus a single dose of polycap for 8 weeks; efficacy to lower blood pressure and elevated lipids and safety assessed as difference with tolerance to double dose of polycap compared to a single dose.
Time Frame: 8 weeks
Measure: Mean (95% Confidence Interval); unit: mmHG
Arm/Group | Two Doses of Low Strength Polycap | One Dose of Low Srength Polycap
Number analyzed (Participants) | 257 | 261
mmHG | 126.6 [122.4 to 132.6] | 129.9 [127.5 to 131.6]

2. Primary Outcome: Tolerability of a Double Dose of Half Strength Polycap
Time Frame: 8 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Blood Pressure Reduction and Lipid Lowering in Type 2 Diabetics
Time Frame: 8 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Two Doses of Low Strength Polycap | One Dose of Low Srength Polycap
Serious Adverse Events (participants affected / at risk) | 9/257 | 1/261
Other Adverse Events (participants affected / at risk) | 5/257 | 4/261
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Two Doses of Low Strength Polycap (N=257) | One Dose of Low Srength Polycap (N=261)
GASTRITIS (Gastrointestinal disorders) | 9 (9) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Two Doses of Low Strength Polycap (N=257) | One Dose of Low Srength Polycap (N=261)
Dry cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No